CLINICAL TRIAL: NCT05700266
Title: Anticoagulation Using Rivaroxaban on Top of Aspirin in Recent Stroke/Transient Ischemic Attack Patients With Intracranial Atherosclerotic Stenosis (AA-ICAS)
Brief Title: Anticoagulation Using Rivaroxaban on Top of Aspirin in Intracranial Atherosclerotic Stenosis
Acronym: AA-ICAS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Kezhong Zhang, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AA-ICAS
Record Dates: First submitted 2022-12-26; First posted 2023-01-26 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Ischemic Stroke; Intracranial Atherosclerosis; Stenosis
Keywords: rivaroxaban, stroke, intracranial atherosclerosis stenosis
MeSH Terms: conditions — Ischemic Stroke; Intracranial Arteriosclerosis; Constriction, Pathologic; Stroke | interventions — Rivaroxaban; Clopidogrel; Aspirin

STUDY DESIGN:
Intervention Model Description: This study is an investigator initiated, randomized, blinded endpoint assessment, clinical trial and conducted at 10 sites in the China. Patients meeting the enrollment criteria will be randomly assigned to one of the two treatment groups (1:1) and will be followed up for 1 year.
Who Masked: Outcomes Assessor
Masking Description: Endpoint assessments, including neurological function evaluation, primary and secondary ending points, will be performed blindly by an assessment group who are blind to this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban and Aspirin (Experimental): Rivaroxaban (2.5mg orally twice a day for 90 days) and Aspirin (100mg once a day for 1 year)
  Interventions: Drug: Rivaroxaban; Drug: Aspirin; Other: Risk Factor Management in both arms
- Clopidogrel and Aspirin (Active Comparator): Clopidogrel (300mg loading dose, then 75mg once daily for 90 days) and Aspirin (100mg once a day for 1 year)
  Interventions: Drug: Clopidogrel; Drug: Aspirin; Other: Risk Factor Management in both arms

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban (2.5mg orally twice a day for 90 days)
  Arms: Rivaroxaban and Aspirin
Drug: Clopidogrel — Clopidogrel (300mg loading dose, then 75mg once daily for 90 days)
  Arms: Clopidogrel and Aspirin
Drug: Aspirin — Aspirin (100mg once a day for 1 year)
Other: Risk Factor Management in both arms — Risk factors for stroke (LDL, blood pressure, non-HDL cholesterol, diabetes, smoking, weight, and physical activity) will be monitored and managed

SUMMARY:
The primary goal of the clinical trial is to test the effect of oral rivaroxaban plus aspirin in patients with recent stroke/ transient ischemic attack (TIA) caused by intracranial artery stenosis. Participants will be divided into 2 groups to receive either oral rivaroxaban plus aspirin or oral clopidogrel plus aspirin. The main question it aims to answer is whether the experimental group (oral rivaroxaban plus aspirin) is superior to the control group ( oral clopidogrel plus aspirin) to lower recurrent stroke/TIA or death in these patients during 1 year of follow-up.

DETAILED DESCRIPTION:
Intracranial atherosclerotic stenosis (ICAS) accounts for up to 30-50% of strokes amongst Asian patient cohorts, in contrast to 5-10% of strokes amongst western patient cohorts. The SAMMPRIS established aggressive medical management (dual antiplatelet therapy using asprin and clopidogrel, intensive management of vascular risk factors, and lifestyle modification) as a superior choice for symptomatic ICAS compared to the percutaneous transluminal angioplasty and stenting. However, around 15% still had recurrent stroke or death during a median follow-up of 32.4 months in SAMMPRIS study in the aggressive medical management group.

Rivaroxaban is a Non-vitamin K antagonist oral anticoagulant (NOAC) that Directly and selectively inhibits factor Xa. 2019 European Society of Cardiology (ESC) recommended that adding rivaroxaban (2.5mg twice a day) to aspirin for long-term secondary prevention in patients with chronic coronary syndromes (post-myocardial infarction >1 year) may be considered (IIB). 2020 ESC also recommended the adding of rivaroxaban (2.5mg twice a day for 1 year) to aspirin plus clopidogrel in acute coronary syndrome (IIB).

The proposed study will directly compare rivaroxaban on top of aspirin with clopidogrel on top of asprin for preventing recurrent stroke/TIA and death in recent stroke/TIA patients with ICAS.

The investigators calculated that a sample of 1180 patients (590 in each arm) would provide 80% power to detect a relative risk reduction of 35% in the ravaxaban-aspirin group, with a two-sided type I error of 0.05, assuming an event rate of 15% in the clopidogrel-aspirin group and a 5% overall rate of withdrawal.

Baseline features of the two groups were compared with the use of an independent group t-test (for means) or chi-square test (for percentages). Analysis of primary and secondary outcomes was based on Kaplan-Meier estimates of cumulative incidence. All analyses were performed on an intention-to-treat basis, unless specified otherwise. All tests were two-sided, and a P value of 0.05 was considered to indicate statistical significance. All statistical analyses were performed with the use of SPSS software.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 30 years and ≤ 75 years
2. TIA or Acute ischemic stroke that occurred within 30 days prior to randomization.
3. Modified Rankin score of ≤ 3
4. TIA or Acute ischemic stroke attributed to a 50 to 99% stenosis of a major intracranial artery (internal carotid artery [ICA], vertebral artery [VA], basilar artery [BA] and the M1 segment of middle cerebral artery [MCA]). The diagnostic evaluation for ICAS at each site is confirmed by the local investigator, using magnetic resonance angiography (MRA), or computerized tomographic angiography (CTA), high resolution MR, or digital substraction angiography (DSA).
5. To increase the likelihood that the symptomatic intracranial stenosis is atherosclerotic, patients aged 30-49 years are required to meet at least one additional criteria (i-vi) below:

   i. insulin dependent diabetes for at least 15 years. ii. at least 2 of the following atherosclerotic risk factors: hypertension (blood pressure ≥ 140/90 or on antihypertensive therapy); dyslipidemia (low density lipoprotein [LDL] ≥ 130 mg /dl or high density lipoprotein [HDL] < 40 mg/dl or fasting triglycerides ≥150 mg/dl or on lipid lowering therapy); smoking; non-insulin dependent diabetes or insulin dependent diabetes of less than 15 years duration; family history of any of the following: myocardial infarction, coronary artery bypass, coronary angioplasty or stenting, stroke, carotid endarterectomy or stenting, peripheral vascular surgery in parent or sibling who was < 55 years of age for men or < 65 for women at the time of the event.

   iii. history of any of the following: myocardial infarction, coronary artery bypass, coronary angioplasty or stenting, carotid endarterectomy or stenting, or peripheral vascular surgery for atherosclerotic disease.

   iv. any stenosis of an extracranial carotid or vertebral artery, another intracranial artery, subclavian artery, coronary artery, iliac or femoral artery, other lower or upper extremity artery, mesenteric artery, or renal artery that was documented by non-invasive vascular imaging or catheter angiography and is considered atherosclerotic. v. aortic arch atheroma documented by non-invasive vascular imaging or catheter angiography.

   vi. any aortic aneurysm documented by non-invasive vascular imaging or catheter angiography that is considered atherosclerotic.
6. Patient agrees with follow-up visits and is available by phone.
7. Patient understands the purpose and requirements of the study, can make him/herself understood, and has signed informed consent.

Exclusion Criteria:

1. Previous treatment of target intracranial lesion with a stent, angioplasty, or other mechanical devices (e.g. mechanical thrombectomy, coil embolization)
2. Plan to perform angioplasty, stenting, coiling, thrombectomy, endarterectomy or aneurysmal coil embolization for any other cerebral blood vessels (common carotid artery [CCA], ICA, VA, MCA, anterior cerebral artery [ACA], posterior cerebral artery [PCA] et al)
3. Intracranial tumor (except meningioma) or any intracranial vascular malformation
4. Thrombolytic therapy within 24 hours prior to randomization
5. Progressive neurological signs within 24 hours prior to enrollment
6. History of any intracranial hemorrhage (parenchymal, subarachnoid, subdural, epidural)
7. Intracranial arterial stenosis due to arterial dissection; MoyaMoya disease; any known vasculitic disease; viral vasculopathy; neurosyphilis; any other intracranial infection; any intracranial stenosis associated with cerebral spinal fluid pleocytosis; radiation induced vasculopathy; fibromuscular dysplasia; sickle cell disease; neurofibromatosis; benign angiopathy of central nervous system; postpartum angiopathy; suspected vasospastic process; reversible cerebral vasoconstriction syndrome (RCVS); suspected recanalized embolus
8. Presence of any of the following unequivocal cardiac sources of embolism: chronic or paroxysmal atrial fibrillation, mitral stenosis, mechanical valve, endocarditis, intracardiac clot or vegetation, myocardial infarction within three months, dilated cardiomyopathy, left atrial spontaneous echo contrast, ejection fraction less than 30%
9. Known allergy or contraindication to aspirin, clopidogrel or rivaroxaban.
10. Active peptic ulcer disease, major systemic hemorrhage within 30 days, active bleeding diathesis, platelets < 100,000, hematocrit < 30, international normalized ration [INR] > 1.5, clotting factor abnormality that increases the risk of bleeding, current alcohol or substance abuse, uncontrolled severe hypertension (systolic pressure > 180 mm Hg or diastolic pressure > 115 mm Hg), severe liver impairment (aspartate transaminase [AST] or alanine transaminase [ALT] > 3 x normal, cirrhosis), creatinine > 3.0 (unless on dialysis)
11. Major surgery (including open femoral, aortic, cardiac or carotid surgery) within previous 30 days or planned in the next 1 year after enrollment.
12. Any condition other than intracranial arterial stenosis that requires the subject to take any antithrombotic medication other than aspirin (NOTE: exceptions allowed for use of subcutaneous heparin for deep vein thrombosis (DVT) prophylaxis while hospitalized)
13. Severe neurological deficit that renders the patient incapable of living independently
14. Dementia or psychiatric problem that prevents the patient from relevant evaluation or follow-up reliably
15. Co-morbid conditions that may limit survival to less than 1 year
16. Currently breastfeeding, pregnancy or of childbearing potential and unwilling to use contraception for the duration of this study
17. Enrollment in another study that would conflict with the current study.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1180 (Estimated)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
any stroke (ischemic or hemorrhagic) or death during 1 year of follow-up | the primary outcome will be assessed during 1 year of follow-up after recruitments.

SECONDARY OUTCOMES:
Changes in the neurological function recovery | Neurological function will be evaluated at 90 days, 6 months and 1 year after recruitments.
  Neurological function will be evaluated using National Institute of Health stroke scale (NIHSS), modified Ranking Scale.
Major non-intracranial bleeding | during 1 year of follow-up after recruitments.
  Major non-intracranial bleeding is defined according to the International Society on Thrombosis and Haemostasis (ISTH) criteria:
  clinically overt bleeding with a fatal outcome, a reduction in haemoglobin level of ≥20 g/l within 7 days, transfusion of at least two units of blood, or symptomatic bleeding in a critical area or organ (intraspinal, intraocular, pericardial, intra-articular, intramuscular with compartment syndrome, retroperitoneal).
Clinically relevant non-major bleeding | during 1 year of follow-up after recruitments.
  Clinically relevant non-major bleeding is defined as bleeding not fulfilling the ISTH criteria, but that was clinically overt and led to hospitalization, change of antithrombotic therapy, or necessitated a medical or surgical intervention.
acute myocardial infarction,acute limb ischemia | during 1 year of follow-up after recruitments.

CONTACTS AND LOCATIONS:
Overall Officials: Kezhong Zhang, Doctor, Study Chair — The First Affiliated Hospital with Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be available to other researchers under reasonable request and approved by the ethics committee.